CLINICAL TRIAL: NCT06660641
Title: TaurolockTMHep100 Versus Saline 0.9% As Secondary Prevention of Catheter-related Bloodstream Infections (CRBSI); a Single Center, Double Blinded, Randomized, Controlled Study in Patients with Chronic Intestinal Failure Dependent on Home Parenteral Support (HPS)
Brief Title: Clinical Trial Comparing TaurolockTMHep100 (Taurolidine 1.35%) and 0.9% Saline As Prevention of Recurrent Catheter-related Bloodstream Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TauroPharm (Industry)
Responsible Party: Principal Investigator, Palle Bekker Jeppesen, MD, PhD, DMSc, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-19000051
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2019-04

CONDITIONS: Catheter Related Blood Stream Infections; Intestinal Failure
Keywords: Taurolidine; Catheter-related bloodstream infections; Intestinal failure
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TaurolockTMHep100 (Active Comparator)
  Interventions: Device: TaurolockTMHep100
- 0.9% saline (Placebo Comparator)
  Interventions: Device: 0.9 % saline

INTERVENTIONS:
Device: TaurolockTMHep100 — 1.35% taurolidine containing catheter losk solution
  Arms: TaurolockTMHep100
Device: 0.9 % saline — placebo
  Arms: 0.9% saline

SUMMARY:
The purpose of the trial is to compare two catheter lock solutions (active: 1.35% taurolidine and placebo: 0.9% saline), on the occurence of catheter related blood stream infection, in patients with intestinal failure and a central venous catheter for home parenteral support.

DETAILED DESCRIPTION:
Patients with long-term intestinal failure rely on Home Parenteral support (HPS) delivered through a central venous catheter(CVC). Catheter Related Blood Stream Infections(CRBSI) are a frequent complication leading to increased morbidity, hospital admissions, cost, and risk of repeated replacement of the CVC. The infections often originate from contamination of the catheter hub, and growth of microorganisms on the inner lumen of the catheter imbedded in a biofilm. To prevent infections good hygiene guidelines and the use of a catheter lock solution is applied.

The primary objective is to compare two catheter lock solutions, 1,35% taurolidine and 0.9% saline, on the occurence of recurrent CRBSIs. The secondary objectives are to compare the two devices according to other catheter-related complications, adverse events and costs.

Patients with at least one prior CRBSI is included. Patients instill the solution in their CVC after each infusion of HPS, with a minimum of three times per week, depending on their individual HPS programme.

Before the blinded randomization the patients will be paired according to age and stratified according to prior CRBSI incidence.

Duration of the instillation will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving HPS at the department of Medical gastroenterology, Rigshospitalet, who have at least one prior CRBSI and thereby demonstrated susceptibility towards developing CRBSI while on HPS and the following:

1. Signed informed consent form
2. Has a single-lumen subcutaneously tunneled CVC
3. Has been at least 3 weeks since termination of the antibiotic treatment for their last CRBSI

Exclusion Criteria:

Patients who:

1. have a known hypersensitivity/allergy to TauroLockTMHep 100 or heparin and/or their excipients
2. are pregnant, lactating or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrent catheter-related bloodstream infections | Treatment time 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nerstrom CT, Scheike T, Moser CE, Tribler S, Jeppesen PB. Taurolidine lock reduces recurrent catheter-related bloodstream infections in patients with chronic intestinal failure: A randomized, placebo-controlled trial in a real-world clinical setting. Clin Nutr. 2025 Aug;51:90-100. doi: 10.1016/j.clnu.2025.05.020. Epub 2025 Jun 3. PMID 40554263